CLINICAL TRIAL: NCT04666870
Title: Shanghai Guanghua Integrated Traditional Chinese and Western Medicine Hospital, Guanghua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, China
Brief Title: Axis Length and Its Relationship With Refractive Error in Chinese University Students
Status: Completed | Type: Observational
Sponsor: Wang Hongxia (Other)
Collaborators: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Wang Hongxia, Shanghai Guanghua Integrated Traditional Chinese and Western Medicine Hospital, Guanghua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine
Organization: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Other Study IDs: 2020-K-106
Record Dates: First submitted 2020-11-02; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Refractive Error - Myopia Axial
Keywords: China; high myopia; hyperopia; emmetropia
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- axis length: 1007 healthy students with moderate to high myopia (SE ≤ -4.00D) and 894 without myopia (-0.50D ≤ spherical power ≤ +2.00D) were enrolled.
  Interventions: Other: myopia or not myopia
- gender: male were 54.29% (N=1032), and female were 45.71% (N=869)
  Interventions: Other: myopia or not myopia

INTERVENTIONS:
Other: myopia or not myopia — visual acuity, IOL master biometry, the anterior segment with slit lamp, dilated fundus examination and refraction.

SUMMARY:
To investigate the relationship between axis length (AL) and refractive error. eyes of low hyperopia to emmetropia subjects, comprising eyes with moderate to high myopia (-11.00D ≤ SE ≤ -4.00D) were analyzed in this cross-sectional study. Cycloplegic refractive error was measured with the autorefractor, AL was measured with the IOL master. Association between AL and refractive error were evaluated by linear regression analysis. The mean of AL and its correlation with SE, sex, and age were evaluated.

DETAILED DESCRIPTION:
To investigate the relationship between axis length (AL) and refractive error (RE). 894 eyes with low hyperopia to emmetropia (-0.50D ≤ spherical equivalent (SE) ≤ +2.00D), comprising 1007 eyes with moderate to high myopia (-11.00D ≤ SE ≤ -4.00D) were analyzed in this study. Cycloplegic RE was measured with the autorefractor, AL was measured with the IOL master. Association between AL and refractive error were evaluated by linear regression analysis. The mean of AL and its correlation with SE, sex, and age were evaluated.

ELIGIBILITY:
Inclusion Criteria:

with moderate to high myopia (SE ≤ -4.00D) without myopia (-0.50D ≤ spherical power ≤ +2.00D) no concurrent eye disease best corrected visual acuity is 1.0

Exclusion Criteria:

significant systemic illnesses congenital myopia, media opacity uveitis glaucoma intraocular surgery refractive surgery neurologic diseases retinal disease

Ages: 22 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The subject recruited for the study were 1935 students
Sampling Method: Probability Sample
Enrollment: 1901 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-11 (Actual)

PRIMARY OUTCOMES:
Axis length | from baseline at 6 months
  Axis length change from baseline at 6 months
Refractive Error | from baseline at 6 months
  Refractive Error change from baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, director, Study Director — Shanghai Guanghua integrated traditional Chinese and Western Medicine Hospital
Locations (1):
- Shanghai Guanghua Integrated Traditional Chinese and Western Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Holden BA, Fricke TR, Wilson DA, Jong M, Naidoo KS, Sankaridurg P, Wong TY, Naduvilath TJ, Resnikoff S. Global Prevalence of Myopia and High Myopia and Temporal Trends from 2000 through 2050. Ophthalmology. 2016 May;123(5):1036-42. doi: 10.1016/j.ophtha.2016.01.006. Epub 2016 Feb 11. PMID 26875007
- [Result] Kempen JH, Mitchell P, Lee KE, Tielsch JM, Broman AT, Taylor HR, Ikram MK, Congdon NG, O'Colmain BJ; Eye Diseases Prevalence Research Group. The prevalence of refractive errors among adults in the United States, Western Europe, and Australia. Arch Ophthalmol. 2004 Apr;122(4):495-505. doi: 10.1001/archopht.122.4.495. PMID 15078666
- [Result] Morgan IG, Ohno-Matsui K, Saw SM. Myopia. Lancet. 2012 May 5;379(9827):1739-48. doi: 10.1016/S0140-6736(12)60272-4. PMID 22559900
- [Result] Mountjoy E, Davies NM, Plotnikov D, Smith GD, Rodriguez S, Williams CE, Guggenheim JA, Atan D. Education and myopia: assessing the direction of causality by mendelian randomisation. BMJ. 2018 Jun 6;361:k2022. doi: 10.1136/bmj.k2022. PMID 29875094
- [Result] Dolgin E. The myopia boom. Nature. 2015 Mar 19;519(7543):276-8. doi: 10.1038/519276a. No abstract available. PMID 25788077
- [Result] Spillmann L. Stopping the rise of myopia in Asia. Graefes Arch Clin Exp Ophthalmol. 2020 May;258(5):943-959. doi: 10.1007/s00417-019-04555-0. Epub 2019 Dec 23. PMID 31873785
- [Result] Battersby K, Koy L, Phillips N, Sim J, Wilk J, Schmid KL. Analysis of physical activity in emmetropic and myopic university students during semester and holiday periods: a pilot study. Clin Exp Optom. 2015 Nov;98(6):547-54. doi: 10.1111/cxo.12327. PMID 26769178
- [Result] Tideman JWL, Polling JR, Jaddoe VWV, Vingerling JR, Klaver CCW. Growth in foetal life, infancy, and early childhood and the association with ocular biometry. Ophthalmic Physiol Opt. 2019 Jul;39(4):245-252. doi: 10.1111/opo.12630. PMID 31236981
- [Result] Jonas JB, Ohno-Matsui K, Panda-Jonas S. Myopia: Anatomic Changes and Consequences for Its Etiology. Asia Pac J Ophthalmol (Phila). 2019 Sep-Oct;8(5):355-359. doi: 10.1097/01.APO.0000578944.25956.8b. PMID 31425168
- [Result] Ohno-Matsui K, Lai TY, Lai CC, Cheung CM. Updates of pathologic myopia. Prog Retin Eye Res. 2016 May;52:156-87. doi: 10.1016/j.preteyeres.2015.12.001. Epub 2016 Jan 6. PMID 26769165
- [Result] Paluru P, Ronan SM, Heon E, Devoto M, Wildenberg SC, Scavello G, Holleschau A, Makitie O, Cole WG, King RA, Young TL. New locus for autosomal dominant high myopia maps to the long arm of chromosome 17. Invest Ophthalmol Vis Sci. 2003 May;44(5):1830-6. doi: 10.1167/iovs.02-0697. PMID 12714612
- [Result] Wang J, Ying GS, Fu X, Zhang R, Meng J, Gu F, Li J. Prevalence of myopia and vision impairment in school students in Eastern China. BMC Ophthalmol. 2020 Jan 2;20(1):2. doi: 10.1186/s12886-019-1281-0. PMID 31898504
- [Result] Richter GM, Wang M, Jiang X, Wu S, Wang D, Torres M, Choudhury F, Varma R; Chinese American Eye Study Group. Ocular Determinants of Refractive Error and Its Age- and Sex-Related Variations in the Chinese American Eye Study. JAMA Ophthalmol. 2017 Jul 1;135(7):724-732. doi: 10.1001/jamaophthalmol.2017.1176. PMID 28520882
- [Result] Rozema JJ, Sun W, Wu JF, Jiang WJ, Wu H, Lu TL, Hu YY, Chen R, Guo DD, Wang XR, Dankert S, Jonas JB, Iribarren R, Tian QM, Bi HS. Differences in ocular biometry between urban and rural children matched by refractive error: the Shandong Children Eye Study. Ophthalmic Physiol Opt. 2019 Nov;39(6):451-458. doi: 10.1111/opo.12649. PMID 31696541
- [Result] Mallen EA, Gammoh Y, Al-Bdour M, Sayegh FN. Refractive error and ocular biometry in Jordanian adults. Ophthalmic Physiol Opt. 2005 Jul;25(4):302-9. doi: 10.1111/j.1475-1313.2005.00306.x. PMID 15953114
- [Result] Zadnik K, Mutti DO, Mitchell GL, Jones LA, Burr D, Moeschberger ML. Normal eye growth in emmetropic schoolchildren. Optom Vis Sci. 2004 Nov;81(11):819-28. doi: 10.1097/01.opx.0000145028.53923.67. PMID 15545807